CLINICAL TRIAL: NCT06518239
Title: Establishing Optimal PEEP Setting for Obese Patients in the Steep Trendelenburg Position: a Pilot Study.
Brief Title: Establishing Optimal PEEP Setting for Obese Patients in the Steep Trendelenburg Position
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Tinashe Maduke (Other)
Responsible Party: Sponsor-Investigator, Tinashe Maduke, Assistant Professor of Medicine, University of Missouri-Columbia
Organization: University of Missouri-Columbia (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2103228
Record Dates: First submitted 2024-06-12; First posted 2024-07-24 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Obesity
Keywords: obesity; steep trendelenburg; Trendelenburg; PEEP; positive end-expiratory pressure; EIT; electrical impedance tomography
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Patients will be monitored by the standard of care anesthesia machines intraoperatively. An EIT belt will be attached to the patient intraoperatively, and data from the belt will be compared to the anesthesia machines.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- PEEP Belt (Experimental): PEEP belt will be placed on the patient intraoperatively. All patients will be monitored using anesthesia machines as standard of care.
  Interventions: Device: Peep Belt

INTERVENTIONS:
Device: Peep Belt — Belt will be placed on the nipple line of the patient prior to the surgery start in the operating room. Data will be collected prior to the initial incision after the patient has been intubated, and then at the end of surgery before the patient has been extubated.
  Other Names: EIT belt; electrical impedance tomography

SUMMARY:
The purpose of this study is to determine whether the Enlight 2100 electrical impedance tomography (EIT) belt can optimize positive end-expiratory pressure (PEEP) during surgery better than standard anesthesia machines.

DETAILED DESCRIPTION:
Positive end-expiratory pressure (PEEP) is a measure taken intraoperatively to manage breathing during surgery. The Enlight 2100 is a device that uses electrical impedance tomography (EIT) to measure PEEP and provide a live image of the lungs while a patient is mechanically ventilated. In this study, the investigators will use the Enlight 2100 EIT belt to measure PEEP intraoperatively in order to better optimize PEEP settings for difficult cases.

ELIGIBILITY:
Inclusion Criteria:

1. BMI ≥ 40 kg/m2
2. Age > 18 years
3. Scheduled for elective laparoscopic abdominal surgery in the steep Trendelenburg position.
4. Able to provide informed consent.

Exclusion Criteria:

1. Currently pregnant.
2. Presence of pacemaker, neurostimulator, spinal cord stimulator, or implantable cardioverter-defibrillator.
3. Skin ulcerations on upper torso near the belt placement.
4. Presence of phrenic nerve palsy or other diaphragm conditions.
5. Thoracic circumference > 134 cm.
6. Tracheomalacia.
7. Inability to speak and understand English.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Optimal PEEP | From the time of consent to the end of surgery, assessed up to 24 hours.
  Optimal positive end-expiratory pressure (PEEP) measured using the electrical impedance tomography (EIT) belt during surgery.

SECONDARY OUTCOMES:
Difference between EIT and standard of care measured PEEP | From the time of consent to the end of surgery, assessed up to 24 hours.
  Measured difference between optimal positive end-expiratory pressure from the study device and the standard of care anesthesia machines.
Delays in extubation | From the day of surgery to discharge, up to 1 week
  Number of delays in extubating the patient due to breathing complications during surgery.
Incidence of extubation complications | From the day of surgery to discharge, up to 1 week
  Number of reintubations needed and/or failed extubations after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Tinashe Maduke, MD, MPH, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University Hospital, Columbia, Missouri, United States